CLINICAL TRIAL: NCT00990574
Title: Spinal Anesthesia for Cesarean Delivery: The Wiley Spinal Catheter Intermittent Bolus Technique Versus Single Shot Spinal Anesthesia
Brief Title: A Study Comparing Two Spinal Techniques for for Cesarean Delivery Anesthesia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: device not found to be adequate
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Brendan Carvalho, Associate Professor of Anesthesia, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SU-10012009-4120; 17492
Record Dates: First submitted 2009-10-05; First posted 2009-10-07 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Hypotension; Headache
MeSH Terms: conditions — Hypotension; Headache

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- spinal anesthesia group (SAG) (Active Comparator): Participants will undergo the standard procedures involved in placement of a spinal anesthetic in the sitting position.
  Interventions: Device: Spinal Anesthesia Group (SAG)
- The WSCG (wiley spinal catheter group) (Active Comparator): The WSCG (wiley spinal catheter group) will undergo the standard procedures involved in placement of a spinal anesthetic in the sitting position.
  Interventions: Device: Wiley Spinal Catheter

INTERVENTIONS:
Device: Wiley Spinal Catheter — The WSCG (wiley spinal catheter group) will have a Wiley spinal catheter placed, but it will not be dosed until the patient is in the supine position with left uterine displacement. Participants will receive the medication (12 mg of 0.75% hyperbaric bupivacaine, 10 mcg of fentanyl, and 100 mcg of morphine) in sequential doses.
  Arms: The WSCG (wiley spinal catheter group)
Device: Spinal Anesthesia Group (SAG) — The SAG (spinal anesthesia group) will have their drugs (12 mg of 0.75% hyperbaric bupivacaine, 10 mcg of fentanyl, and 100 mcg of morphine) dosed intrathecally as a "single shot" while still in the sitting position.
  Arms: spinal anesthesia group (SAG)

SUMMARY:
The purpose of this study is to compare single shot versus sequential bolus spinal technique via a catheter in patients undergoing Cesarean Section. We aim to determine which technique results in less blood pressure reduction and subsequent vasopressor use.

Other study endpoints include the incidence of maternal post dural puncture headaches and nausea and vomiting. In addition blood and CSF will be collected to see if biochemical mediators are related to wound hyperalgesia and healing.

DETAILED DESCRIPTION:
Following IRB approval, the investigators plan to enroll 60 pregnant women (30 in the spinal anesthesia group (SAG), and 30 patients in the Wiley spinal catheter group (WSCG)) undergoing cesarean delivery. Patients will be randomly assigned to one of these two groups.

Both groups will undergo the standard procedures involved in placement of a spinal anesthetic in the sitting position. The SAG will have their drugs dosed intrathecally as a "single shot" while still in the sitting position. The WSCG will have a Wiley spinal catheter placed, but it will not be dosed until the patient is in the supine position with left uterine displacement. Both groups will be dosed with 12 mg of 0.75% hyperbaric bupivacaine, 10 mcg of fentanyl, and 100 mcg of morphine. While the SAG will receive their total dose as a one time bolus, the WSCG patients will receive the medication in sequential doses.

Blood pressure will be monitored every minute after spinal medication is administered until delivery of the baby. Thereafter, it will be monitored at least every 3 minutes. Any blood pressure below 90, 80 and 70% of baseline will be treated with 50, 100 and 150 mcg of phenylephrine, respectively.

In the WSC group, cerebrospinal fluid (CSF) will be collected prior to intrathecal dosing, and then 1 and 5 hours post-spinal utilizing a three-way stopcock incorporated into the IT catheter.

All CSF samples will be analyzed for various nociceptive and inflammatory biochemical mediators using a multiplex bead array immunoassay plate. Venous blood will be drawn prior to spinal dosing and 5 hours afterwards to measure the same cytokines and biochemical mediators.

Participants will be followed for 2 days post cesarean section to monitor for episodes of a spinal or post dural puncture headache (PDPH). A PDPH is defined as an occipital or frontal headache brought on by the erect posture and relieved when the supine posture is assumed. If the PDPH persists longer than 24 h with the same severity, an epidural blood patch (EBP) will be performed. The decision to perform an EBP will always be made by a staff anesthesiologist. Headaches will be monitored daily for 3 days, then at 1 week. Patients will be treated for their headaches per standard methods by an anesthesiologist not involved in the study.

Postoperative pain will be recorded at rest and sitting at 1, 5, 24, 48h post-cesarean using a VPS 0-10 (0=no pain, 10=worse pain imaginable) measure. The area of secondary hyperalgesia surrounding the wound will be measured at 48hours with a von Frey filament. A color laser Doppler will also be used to assess vascular perfusion of the wound 48 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Class I, II patients
* 18-45 year of age
* Uncomplicated singleton, term pregnancy
* Scheduled for Cesarean section

Exclusion Criteria:

* ASA class 3 and above
* Morbid obesity (BMI>40 kg/m2)
* Postpartum tubal ligation after cesarean
* Hypersensitivity and/or prior reaction to opioids
* Ineffective spinal
* Conversion to general anesthesia
* Multiple gestation pregnancy
* Emergency C-section
* Contraindication to regional anesthesia
* History of chronic opioid use

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Blood pressure maintenance | Spinal to End Surgery
Vasopressor use | Spinal to End Surgery

SECONDARY OUTCOMES:
Post-spinal Headache | 1 week
Postoperative pain, wound hyperalgesia and perfusion | 48 h
CSF and blood biochemical nociceptive and inflammatory mediators | 5 h

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Carvalho, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States